CLINICAL TRIAL: NCT06383923
Title: Risk Factors, Prognosis and Prediction Models for Placenta Accreta Without Prior Cesarean Section：A Prospective Cohort Study
Brief Title: Risk Factors, Prognosis and Prediction Models for Placenta Accreta Without Prior Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYSYDL2022015
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-01

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — placenta and uterus
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women: pregnant women without prior cesarean section（CS） who had prenatal check-ups and gave birth at the Obstetrics Department of Peking University Third Hospital from January 1, 2023 to December 31, 2024.

SUMMARY:
1. Identify the risk factors for Placenta accreta spectrum (PAS) disorders in women without prior caesarean section (CS).
2. Clarify the prognostic factors of the disease and explore individualized treatment options to improve the prognosis of patients with this type of disease;
3. Use the cohort's biological sample database to conduct serology, cytology, and histology studies to explore the abnormal uterine immune microenvironment and the impact on uterine spiral artery remodeling in non-scar uterine-placenta accreta disease.

DETAILED DESCRIPTION:
The placenta accreta spectrum (PAS) is defined as abnormal placental trophoblast adherence with a wide range of myometrial invasion. It is a serious pregnancy complication that can lead to severe postpartum hemorrhage, which may necessitate hysterectomy, and could ultimately lead to maternal death.Previous studies have shown that women with the highest risk of PAS disorders are those with a prior cesarean section (CS) who present in the second trimester of pregnancy with any degree of placenta previa or low-lying placenta.PAS patients without prior CS represent about one-third of the entire PAS population.The strategy to identify at-risk patients without a prior CS has yet to be defined. This may lead to under identification of PAS patients without prior CS and create a missed opportunity to plan the delivery and improve prognosis in these women. Established risk factors distinct from prior CS delivery include in vitro fertilization (IVF), intrauterine implants, endometritis, uterine artery embolization manual placental removal, uterine malformation, adenomyosis, submucosal fibroids, smoking, maternal weight, maternal age, parity, and multifetal pregnancy. Large clinical studies focusing on PAS disorders in women without prior CS are, indeed, scarce.This study aims to explore the risk factors and prognosis of PAS without a history of cesarean section and try to establish the prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women without prior cesarean section
* Pregnant women who had prenatal check-ups and gave birth at the Obstetrics Department of Peking University Third Hospital from January 1, 2023 to December 31, 2024

Exclusion Criteria:

* Pregnant women who did not terminate pregnancy at the Obstetrics Department of Peking University Third Hospital
* Pregnant women who gave birth at <28 weeks.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will prospectively collect pregnant women without history of cesarean sections who had prenatal check-ups and gave birth at the Obstetrics Department of Peking University Third Hospital from January 1, 2023 to December 31, 2024.
  The prospective study will exclude those who did not terminate pregnancy or gave birth in our hospital and those who gave birth at <28 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Placenta Accreta Spectrum | 2 years
  Clinical diagnosis and classification standards are based on the diagnostic standards recommended by FIGO in 2019

SECONDARY OUTCOMES:
Amount of bleeding | 2 years
  Amount of bleeding in 24 hours after delivery
Hemostatic measures | 2 years
  hemostatic measures after delivery
hysterectomy | 2 years
  hysterectomy during the perinatal period
blood transfusion volume | 2 years
  Postpartum blood transfusion volume

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided